CLINICAL TRIAL: NCT02399345
Title: An Open-Label, Treatment Duration-Ranging Study to Evaluate the Safety and Efficacy of Ombitasvir/Paritaprevir/ Ritonavir (Ombitasvir/ABT-450/r) and Dasabuvir Co-administered With Sofosbuvir (SOF) With and Without Ribavirin (RBV) in Direct-Acting Antiviral Agent (DAA) Treatment-Naive Adults With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection
Brief Title: Ombitasvir/Paritaprevir/Ritonavir and Dasabuvir Co-Administered With Sofosbuvir With and Without Ribavirin in Treatment-Naive HCV Genotype 1-Infected Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-310; 2014-005280-32 (EudraCT Number)
Record Dates: First submitted 2015-03-23; First posted 2015-03-26 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Hepatitis C Virus (HCV Infection Genotype 1)
Keywords: Treatment naive; Hepatitis C Genotype 1
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Viekira Pak; ombitasvir; paritaprevir; dasabuvir; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ombitasvir/Paritaprevir/r, Dasabuvir, and SOF plus RBV (Experimental): Ombitasvir/paritaprevir/ritonavir (ombitasvir/paritaprevir/r) (25 mg/150 mg/100 mg once daily) with dasabuvir (250 mg twice daily) and sofosbuvir (SOF) (400 mg once daily), plus weight-based ribavirin (RBV) (dosed 1,000 or 1,200 mg daily divided twice a day) for 6 weeks.
  Interventions: Drug: ombitasvir/paritaprevir/ritonavir, dasabuvir; Drug: sofosbuvir (SOF); Drug: ribavirin (RBV)

INTERVENTIONS:
Drug: ombitasvir/paritaprevir/ritonavir, dasabuvir — tablet; ABT-450 coformulated with ritonavir and ABT-267, ABT-333 tablet
  Other Names: Viekira PAK; ombitasvir also known as ABT-267; paritaprevir also known as ABT-450; dasabuvir also known as ABT-333
Drug: sofosbuvir (SOF) — tablet
Drug: ribavirin (RBV) — tablet

SUMMARY:
This open-label study will evaluate the safety and efficacy of co-formulated ombitasvir/paritaprevir/ritonavir and dasabuvir co-administered with sofosbuvir with or without ribavirin administered for either 4 or 6 weeks in treatment naive adults with chronic HCV-genotype 1 infection without cirrhosis

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years of age at time of screening
2. Chronic Hepatitis C virus (HCV) infection prior to study enrollment
3. Screening laboratory results from the central clinical laboratory indicating HCV genotype 1 infection only
4. Absence of cirrhosis and advanced bridging fibrosis

Exclusion Criteria:

1. Positive test result for hepatitis B surface antigen (HbsAg) or human immunodeficiency virus (HIV) positive immunoassay
2. Clinically significant abnormalities or co-morbidities, other than HCV infection, that make the subject an unsuitable candidate for this study or treatment with Ribavirin (RBV) in the opinion of the investigator
3. Any current or past clinical evidence of cirrhosis such as ascites or esophageal varices, or prior biopsy showing cirrhosis or advanced bridging fibrosis, e.g., a Metavir score > 2 or an Ishak score > 3
4. Use of medications contraindicated for ombitasvir/paritaprevir/ritonavir, dasabuvir, sofosbuvir, or ribavirin (RBV; for those that receive RBV), within 2 weeks or 10 half-lives whichever is longer, prior to study drug administration
5. Current enrolment in another clinical study, previous enrolment in this study, or previous use of any investigational or commercially available anti-HCV agents

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Cohen, MD, Study Director — AbbVie

REFERENCES:
- See also: Related info. — http://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total 10 participants were enrolled in the first arm (ombitasvir/paritaprevir/r, dasabuvir, and SOF plus RBV for 6 weeks); based on inadequate efficacy in the first arm, subsequent arms (4 weeks of treatment; with or without RBV) were not enrolled per protocol.
Period: Overall Study
Arm/Group | Ombitasvir/Paritaprevir/r, Dasabuvir, and SOF Plus RBV
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ombitasvir/Paritaprevir/r, Dasabuvir, and SOF Plus RBV
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 Weeks (SVR12) Post-treatment
Description: The percentage of participants with sustained virologic response (plasma Hepatitis C virus ribonucleic acid [HCV RNA] level less than the lower limit of quantitation [< LLOQ]) 12 weeks after the last dose of study drug. The LLOQ for the assay was 25 IU/mL.
Time Frame: 12 weeks after the last actual dose of study drug
Population: Intent-to-treat (ITT) population: All randomized participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/r, Dasabuvir, and SOF Plus RBV
Number analyzed (Participants) | 10
percentage of participants | 80

2. Secondary Outcome: Percentage of Subjects With On-treatment Virologic Failure
Description: Virologic failure during treatment was defined as confirmed HCV RNA ≥ LLOQ after HCV RNA < LLOQ during treatment; confirmed increase from nadir in HCV RNA (defined as 2 consecutive HCV RNA measurements > 1 log10 IU/mL above nadir) during treatment; or failure to suppress during treatment (defined as all values of HCV RNA ≥ LLOQ during treatment).
Time Frame: 6 weeks
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/r, Dasabuvir, and SOF Plus RBV
Number analyzed (Participants) | 10
percentage of participants | 0

3. Secondary Outcome: Percentage of Subjects With Post-treatment Relapse
Description: Percentage of subjects with HCV RNA less than the lower limit of quantification at the end of treatment with confirmed HCV RNA greater than or equal to the lower limit of quantification through 12 weeks post treatment
Time Frame: Up to 12 weeks after last actual dose of active study drug
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Ombitasvir/Paritaprevir/r, Dasabuvir, and SOF Plus RBV
Number analyzed (Participants) | 10
percentage of participants | 20

ADVERSE EVENTS:
Time Frame: Treatment-emergent Adverse Events (TEAEs) were collected from first dose of study drug until 30 days after the last dose of study drug (up to 10 weeks); Serious Adverse Events (SAEs) were collected from the time informed consent was obtained (up to 15 weeks).
Arm/Group | Ombitasvir/Paritaprevir/r, Dasabuvir, and SOF Plus RBV
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ombitasvir/Paritaprevir/r, Dasabuvir, and SOF Plus RBV (N=10)
ANXIETY (Psychiatric disorders) | 1
PHYSICAL ASSAULT (Social circumstances) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ombitasvir/Paritaprevir/r, Dasabuvir, and SOF Plus RBV (N=10)
EAR DISCOMFORT (Ear and labyrinth disorders) | 1
DRY EYE (Eye disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 2
FLATULENCE (Gastrointestinal disorders) | 1
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 2
ASTHENIA (General disorders) | 1
CHILLS (General disorders) | 1
FATIGUE (General disorders) | 5
INFLAMMATION (General disorders) | 1
GASTROENTERITIS (Infections and infestations) | 1
ORAL HERPES (Infections and infestations) | 1
TOOTH INFECTION (Infections and infestations) | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 3
VIRAL INFECTION (Infections and infestations) | 1
CONCUSSION (Injury, poisoning and procedural complications) | 1
HAIR INJURY (Injury, poisoning and procedural complications) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1
POLYARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
DIZZINESS (Nervous system disorders) | 1
DYSGEUSIA (Nervous system disorders) | 1
HEADACHE (Nervous system disorders) | 3
MENTAL IMPAIRMENT (Nervous system disorders) | 1
NEURALGIA (Nervous system disorders) | 1
AGORAPHOBIA (Psychiatric disorders) | 1
INSOMNIA (Psychiatric disorders) | 5
IRRITABILITY (Psychiatric disorders) | 2
NIGHTMARE (Psychiatric disorders) | 1
POLLAKIURIA (Renal and urinary disorders) | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 1
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 1
SKIN ATROPHY (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.